CLINICAL TRIAL: NCT01002378
Title: A Phase I, Randomized, Open Label, 3-Way Cross-Over Study to Determine the Effect of a High-Fat Breakfast, a Low-Fat Breakfast and Fasting State on the Pharmacokinetics of a Single Oral Dose of 160 mg Regorafenib (BAY73-4506) in Healthy Volunteers
Brief Title: The Effect of Food (High Fat and Low Fat Breakfast) on the Pharmacokinetics of Regorafenib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare Pharmaceuticals Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 14656
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Dietary Fats; Pharmacokinetics
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Arm 2 (Experimental)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Arm 3 (Experimental)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — A single dose of regorafenib will be administered immediately following a high fat breakfast
  Arms: Arm 1
Drug: Regorafenib (Stivarga, BAY73-4506) — A single dose of regorafenib will be administered immediately following a low fat breakfast
  Arms: Arm 2
Drug: Regorafenib (Stivarga, BAY73-4506) — A single dose of regorafenib will be administered following an overnight fast
  Arms: Arm 3

SUMMARY:
An open label, three way crossover study to determine the effect of a high fat breakfast or a low fat breakfast on the pharmacokinetics of a single dose of regorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 45 years (inclusive) at the first Screening examination
* BMI: between 18 and 32 kg / m²

Exclusion Criteria:

* Regular use of medicines at the time of Screening, including prescription medications, herbal supplements and high dose vitamins
* Sitting systolic BP > 140 mmHg or Diastolic BP > 90 or < 60 mmHg
* History of hypersensitivity or allergy
* History of somatic or psychiatric disease/condition, which may interfere with the objectives of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Primary PK parameters: AUC, Cmax of BAY 73-4506 | Samples up to 336 hours post dose

SECONDARY OUTCOMES:
Sec. PK Parameters: tmax and t1/2 of BAY73-4506 | Samples up to 336 hours post dose
AUC, Cmax, tmax and t1/2 of Metabolites | Samples up to 336 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Brighton, Massachusetts, United States